CLINICAL TRIAL: NCT04451460
Title: Frequency and Effect on the Prognosis of Hyponatremia During the diagnosıs in Small Cell Lung Cancer
Brief Title: Effect of Hyponatremia in Small Cell Lung Cancer
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Other Study IDs: AnkaraSanatoryum
Record Dates: First submitted 2020-06-01; First posted 2020-06-30 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Small Cell Lung Cancer
Keywords: Small cell lung cancer; hyponatremia; prognosis; treatment; biochemistry
MeSH Terms: conditions — Small Cell Lung Carcinoma; Hyponatremia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hyponatremia: Hyponatremic small cell cancer patients
- Normonatremia: Normonatremic small cell cancer patients

SUMMARY:
In this retrospective study, the investigators determined the frequency of hyponatremia in small cell lung cancer and the prognosis. 126 (27%) of 466 patients were hyponatremic. Hyponatremia could not be corrected in 50.8% (n=64) of hyponatremic patients. Survival was found to be better in the group of whom hyponatremia was corrected.

ELIGIBILITY:
Inclusion Criteria:

Patients diagnosed with SCLC between January 2012 and January 2017 in our hospital were retrospectively screened

Exclusion Criteria:

Over 18 age If data doesn't exist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with SCLC between January 2012 and January 2017 in our hospital were retrospectively screened
Sampling Method: Non-Probability Sample
Enrollment: 466 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
Mortality | Through study completion, an average of 3 months
  Effect of hyponatremia according to mortality